CLINICAL TRIAL: NCT03789435
Title: Medium-term Incidence Study of Phantom Limb Syndrome in Trans Femoral and Trans Tibial Amputated Patients
Brief Title: Pain in Trans Femoral and Trans Tibial Amputees
Acronym: AMPUPHANTOM
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Mariagrazia Benedetti, Head Physical Medicine and Rehabilitation Unit, Istituto Ortopedico Rizzoli
Other Study IDs: 0013569
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Lower Limb Amputation Above Knee; Lower Limb Amputation Below Knee
MeSH Terms: interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amputees: Patients underwent trans-tibial and trans-femoral amputation of any etiology at the Rizzoli Orthopedic Institute from 2015 to 2017 with the presence of analgesia data for surgery in a computerized record (SIR, Rizzoli information system). A questionnaire for the detection of residual limb pain will be administrate to all the survivors.
  Interventions: Diagnostic Test: Questionnaire

INTERVENTIONS:
Diagnostic Test: Questionnaire — A questionnaire from which the session dedicated to the evaluation of the stump pain, the phantom limb and the sensation of the phantom limb has been extracted will be administered: this is the Prosthetic Evaluation Questionnaire (PEQ) validated in Italian by Ferrero et al. 2005.
  In the questionnaire sent to patients will be asked also for anthropometric data (weight, height) in addition to the characteristics of the worn prosthesis and if they have followed a period of rehabilitation.The time of use of the prosthesis will be evaluated through the Houghton Scale of Prosthetic Use in People with Lower- Extremity Amputations (19)

SUMMARY:
Phantom limb is difficult to manage and has a significant impact on the patient's quality of life. At present, the scientific evidence shows that the infusion of local anesthetics with epidural and perineural catheters in the perioperative phase correlates with good pain control in the immediate post-operative, expressed in terms of reduced demand for opiates by the patient undergoing amputation. of lower limb. Few are studies that highlight the effectiveness of such treatments in the medium and long-term prevention of phantom limb syndrome.

The study aims to evaluate the incidence in the medium term of the phantom limb in trans femoral and trans tibial amputees and the possible relationship with the use of adequate pre and perioperative analgesia using peridural and peripheral nerve catheters. The results of the study could provide indications about the need to modify both the perioperative analgesic therapy protocol and also rehabilitation for lower limb amputation surgery in order to reduce the prevalence of phantom limb syndrome with consequent improvement in quality of life.

DETAILED DESCRIPTION:
The prevalence of phantom limb varies from 50-90% in amputated patients. When present, it is difficult to manage and has a significant impact on the patient's quality of life. The causes that determine the development and above all the persistence of this remote syndrome are not known, however some studies report the importance of psychological factors, also related to the time of use of the prosthesis.

After an amputation it is possible to have different pictures of residual pain that are classified as:

* Stump pain (residual limb pain -RLP): described as burning, shock, cut, hypersensitivity of the stump (post-surgical nociceptive, neurogenic, protesigenic, arthrogenic, ischemic, sympathetic, from adhesive scar tissue or hetero topical ossifications, has a incidence of 74% and may persist up to 14 years after amputation.
* Phantom limb pain (PLP) pain: described as a similar neuropathic (cutting, traction, shock pain) and as a similar nociceptive (deaf, cramp-like, compressive), is present in the first 6 months after amputation, but can last for years, and affects up to 85% of patients.
* Phantom limb sensations (phantom sensations - PSs): non-painful perceptions from the part of the body lost after deafferentation or amputation (kinetic, kinesthetic and exteroceptive), is common in the postoperative period, in one third of patients within 24 hours , in three quarters of patients within 4 days, and in 90% of patients, persist within 6 months of surgery.

At present, the scientific evidence shows that the infusion of local anesthetics with perioperative epidural and perineural catheters correlates with good pain control in the immediate post-operative period expressed in terms of reduced opiate demand by of the patient undergoing limb amputation. However, there are no studies on the medium to long-term incidence of phantom limb syndrome in patients who have been treated with multimodal analgesic protocols. Only the observational study performed by Borghi et al. showed that a 3% incidence of phantom limb syndrome in patients treated with prolonged infusion for an average of 30 days with a 0.5% ropivacaine perineural catheter was shown 12 months after limb amputation surgery. Based on this experience for years at the Rizzoli Orthopedic Institute, peridural and peripheral catheters are applied with a dedicated protocol. At present, however, there is no further assessment of the incidence of phantom limb in patients amputated to the IOR who have followed the protocols in use.

Aim The study aims to evaluate the incidence of phantom pain in the medium term, the sensation of phantom limb and the pain of the stump in amputated trans femoral and trans tibial patients operated on the IOR who followed the perioperative analgesic protocol with use of catheters peridural and peripheral nerves. The results of the study could provide indications about the need to modify the perioperative and rehabilitative analgesic therapy protocol for lower limb amputation surgery to favor a reduction in the intensity, prevalence and frequency of phantom limb syndrome with consequent improvement in the quality of life.

Methods Administration (post delivery and supervised compilation by telephone) of the Prosthetic Evaluation Questionnaire (PEQ), of the Houghton Scale of Prosthetic Use in People with Lower-Extremity Amputations and collection of general information : presence and severity of the stump pain, phantom limb pain and phantom limb sensation, weight, height, type of prosthesis and time of use, specific rehabilitation for phantom limb, pharmacological therapy in place.

Type of anesthesia used during surgery and general and local analgesic therapy (perinervous or peridural catheters) used will be retrieved from clinical folders.

Timetable Month 1

* Request to the Institute Informatic System of the identification of patient records with amputation above or below the knee in the years 2015-2017
* Search for computerized folders and data collection of anesthesia and analgesia in a database Month 2
* Identification of patients eligible for the study with consultation of the registry for the search for the deceased
* Sending patient questionnaires and phone calls for completion Month 3
* Collection of questionnaires
* Completion of the database
* Statistic analysis

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing trans-tibial and trans-femoral amputation of any etiology at the Rizzoli Orthopedic Institute from 2015 to 2017
* Presence of analgesia data for surgery in a computerized record (SIR, Rizzoli information system)
* Patients who have accepted to join the study

Exclusion criteria:

* Patients with a medical record inaccessible via SIR (not yet digitized)
* Deceased patients
* Patients under the age of 18
* Non-ambulatory patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients amputated above and below the knee at the Orthopedic Divisions of the Rizzoli Orthopedic Institute
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Mid-term incidence (1 to 3 years) of pain in the stump or phantom limb and phantom limb sensation in amputated trans femoral and trans tibial patients treated at IOR from 2015 to 2017. | 7 days
  Data will be obtained by means of questionnaire sent to patients.
Evaluation of the type of anesthesia and perioperative analgesic treatment with peripheral nerve block effected and of the use of the prosthesis to evaluate possible relations with the presence and the entity of the phantom limb. | 7 days
  Anesthesia data will be retrieved from patient records.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Benedetti, Principal Investigator — IRCCS-Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS-Istituto Ortopedico Rizzoli, Bologna, Italy